CLINICAL TRIAL: NCT01409252
Title: Long Term Neurological and Cognitive Outcome After Neurosurgical Operation for Hemorrhagic Stroke (Intracerebral Hemorrhage)
Brief Title: Long Term Outcome After Hemorrhagic Stroke Surgery
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, George KC Wong, Professor (Clinical), Chinese University of Hong Kong
Other Study IDs: GW007
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Stroke
Keywords: Stroke; intracerebral hemorrhage; surgery
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemorrhagic stroke patients

SUMMARY:
The investigators retrospectively reviewed all patients with neurosurgical operations for hemorrhagic stroke (intracerebral hemorrhage) between 1999 and 2008. Research assistant then telephoned the survivors for neurological and cognitive status.

DETAILED DESCRIPTION:
Death at one year for intracerebral hemorrhage varies by location, with 42% for cerebellar in one series. Of patients who had intracerebral hemorrhage in the United States during 2002, only 20% are expected to be functionally independently at 6 months. Although case series established the value of selected timely hematoma evacuation, long term clinical outcome, especially on cognition, is not well described in the literature. With these in mind, we carried out this study.

ELIGIBILITY:
Inclusion Criteria:

* All hemorrhagic stroke patients with neurosurgical operations performed between 1999 and 2008.

Exclusion Criteria:

* Spontaneous subarachnoid hemorrhage as the dominant etiology
* uncommunicable patients
* nonsurvivors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spontaneous intracerebral hemorrhage with neurosurgical operations
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale | Cross-sectional at 2-12 years after ictus

SECONDARY OUTCOMES:
Barthel Index | Cross-sectional at 2-12 years post-ictus
  Basic Activity of Daily Living
Telephone Interview of Cognitive Status | Cross-sectional at 2-12 years post-ictus

CONTACTS AND LOCATIONS:
Overall Officials: George Wong, MD(CUHK) FRCSEd(SN), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Surgery, The Chinese University of Hong Kong, Hong Kong, China